CLINICAL TRIAL: NCT06613529
Title: Effectiveness of Online Mindfulness Platform in Improving Anxiety, Depression, and Stress in Adults During the COVID-19 Pandemic: a Randomized Control Trial
Brief Title: Effectiveness of Online Mindfulness Platform in Improving Anxiety, Depression, and Stress in Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: N202207017
Record Dates: First submitted 2024-08-29; First posted 2024-09-26 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-08

CONDITIONS: COVID-19 Pandemic; Emotions; Online Mental Health Program
Keywords: COVID-19, physiology, psychology; Mindfulness; online mindfulness
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- online mindfulness group (Experimental): Patients in the experimental group received online mindfulness interventions at least once a week approximately 15-20 minutes each time.
  Interventions: Other: online mindfulness training

INTERVENTIONS:
Other: online mindfulness training — Use publicly available online mindfulness training resources. The training content was to guide patients to practice mindfulness techniques, including "where the body is, the mind is" and "relaxation learning".

SUMMARY:
During the COVID-19 pandemic, adults may experience emotional stress and impact. To reduce the risk of cross-infection, this study aims to use online mindfulness training to improve emotional well-being during the pandemic and assess their effectiveness.

DETAILED DESCRIPTION:
he COVID-19 pandemic had a detrimental global impact on the health of most populations. It causes and also generates further damage to physiology and psychology. Mindfulness is recognized as an effective method for improving the symptoms of physical and mental problems. The purpose of this review will explore the efficacy of an online mindfulness intervention for individuals or groups that impacted symptoms of physiology and psychology in adults during the pandemic base on the principle of evidence-based medicine. At the same time, a set of mindfulness intervention plans will be developed based on the best evidence searched, and a pilot study will be conducted. Therefore, this research design will be divided into two stages. In the first stage, six electronic bibliographic databases will be comprehensively searched for randomized controlled trials that have been published from February 2020 to currently published articles. The research subjects are adults who live in the community and accept online mindfulness intervention. Quality assessment will be performed according to the Cochrane Collaboration's Risk of Bias tool will be used for randomized controlled clinical trials (RCTs). A meta-analysis of the intervention timing and measurements will be performed using Review Manager 5.1 software. The second phase will be a randomized controlled trial pilot study of mindfulness interventions, The research subjects will be divided into two groups, namely the mindfulness intervention experimental group (E) and the control group (C). The researcher uses structured questionnaires to collect data before intervention (To) and at 4 weeks (T1), 8 weeks (T2) after the intervention. Data will be analyzed using the Generalized Estimating Equation to analyze the repeated measurements and intention-to-treat analysis for reducing attrition bias.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 20 years of age
* Conscious
* Able to communicate in Taiwanese

Exclusion Criteria:

* Patients currently receiving antidepressant or anti-anxiety medications
* Patients unable to communicate verbally
* Patients who refuse to provide informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Assessment of anxiety | Anxiety was assessed before the intervention, and at 4 and 8 weeks after the intervention.
  Anxiety levels were assessed using the odd-numbered questions of the Hospital Anxiety and Depression Scale (HADS-14). The full title of HADS-14 is Hospital Anxiety and Depression Scale. This scale consists of 14 items, with 7 items specifically measuring anxiety, known as the Anxiety Subscale (HADS-A).
  Each item in the Anxiety Subscale is rated on a 4-point Likert scale, ranging from 0 (no symptoms) to 3 (significant symptoms). The total score for the anxiety subscale can range from 0 to 21. Higher scores indicate worse outcomes, specifically reflecting greater levels of anxiety.
  The scoring is categorized as follows:
  * 0-7: Normal anxiety levels
  * 8-10: Borderline abnormal anxiety (suggesting possible anxiety)
  * 11-21: Abnormal anxiety (indicating clinical levels of anxiety)

SECONDARY OUTCOMES:
Assessment of depression | Depression was assessed before the intervention, and at 4 and 8 weeks after the intervention.
  Depression levels were assessed using the even-numbered questions of the Hospital Anxiety and Depression Scale (HADS-14). This scale consists of 14 items, with 7 items specifically measuring depression, known as the The full title of HADS-14 is Hospital Anxiety and Depression Scale. Depression Subscale (HADS-D).
  Each item in the Depression Subscale is rated on a 4-point Likert scale, ranging from 0 (no symptoms) to 3 (significant symptoms). The total score for the depression subscale can range from 0 to 21. Higher scores indicate worse outcomes, specifically reflecting greater levels of depression.
  The scoring is categorized as follows:
  * 0-7: Normal depression levels
  * 8-10: Borderline abnormal depression (suggesting possible depression)
  * 11-21: Abnormal depression (indicating clinical levels of depression)

OTHER OUTCOMES:
Assessment of stress | Stress levels were assessed before the intervention, and at 4 and 8 weeks after the intervention.
  Stress levels were assessed using the Perceived Stress Scale (PSS-10). The full title of PSS-10 is Perceived Stress Scale. This scale consists of 10 items. Each item in the scale is rated on a 5-point Likert scale, ranging from 0 (Never) to 4 (Very Often). The total score ranges from 0 to 40. Higher scores indicate worse outcomes, specifically reflecting a higher perceived level of stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Xinyi District, Taiwan

IPD SHARING:
Plan to Share IPD: No